CLINICAL TRIAL: NCT04815161
Title: ASsessment of Adherence TO Medication in AtRIAl Fibrillation - an eMonitoring Drug Dispensing Device Study
Acronym: ASTORIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Pilloxa (Industry)
Responsible Party: Principal Investigator, Dan Atar, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 171965
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Adherence, Patient; Atrial Fibrillation
MeSH Terms: conditions — Patient Compliance; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilloxa pillbox (Other): Patients receiving the Pilloxa pillbox for drug administration
  Interventions: Behavioral: Adherence

INTERVENTIONS:
Behavioral: Adherence — Adherence to medication using an electronic pillbox

SUMMARY:
The ASTORIA study is a prospective cohort single-armed multicenter observational study that aims to assess adherence to rivaroxaban using a high technological electronical pillbox connected to a phone application in a group of atrial fibrillation patients with indication of long term anticoagulation treatment in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient with age > 18 years
* Patients with atrial fibrillation
* Patients initiated, continued on or switched to rivaroxaban for the indication atrial fibrillation with intended lifelong treatment (CHA2 DS2-VASc score ≥ 1).
* The patient must agree to the use of the electronic medication adherence monitoring device, the so-called Pilloxa box and need to have a sufficient understanding of the app and functionality in conjunction with the use of the Pilloxa box.
* Signed informed consent
* No participation in an investigational program with interventions outside of routine clinical practice
* No contra-indications according to the local marketing authorization

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contra-indications according to the local marketing authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence | 2 years
  The rate of adherence to rivaroxaban in a group of atrial fibrillation patients using the Pilloxa box will be assessed.

SECONDARY OUTCOMES:
Persistence rate | 2 years
  Rate of persistence to rivaroxaban in a group of atrial fibrillation patients using the Pilloxa box will be assessed
Rates of risk factors | 2 years
  Risk factors for non-adherence and non-persistence in these patients will be evaluated
Rates of different patient experiences | 2 years
  Patient experiences with the Pilloxa box and application will be evaluated using questionnaires and quality intervjues

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, MD, PhD, Principal Investigator — Univerity of Oslo, Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.